CLINICAL TRIAL: NCT03095391
Title: A Phase 2b Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of FAST PV and mGFR Technology™ in Healthy Subjects and Patients With Varying Degrees of Renal Impairment
Brief Title: The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of FAST PV and mGFR Technology™
Status: Completed | Type: Observational
Sponsor: FAST BioMedical (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 36770001
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2017-10

CONDITIONS: Kidney Diseases; Renal Insufficiency, Chronic; Acute Kidney Injury; Urologic Diseases; Renal Insufficiency
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Acute Kidney Injury; Urologic Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (4):
- Cohort 1: GFR: ≥ 60 mL/min/1.73 m2 VFI dose: 47 mg/3 mL Number of doses: 1 Comparator: none Comparator dose: none
  Interventions: Device: VFI
- Cohort 2: GFR: ≥ 60 mL/min/1.73 m2 VFI dose: 47 mg/3 mL Number of doses: 2 Comparator: Iohexol 5 mL Comparator dose: 1
  Interventions: Device: VFI; Device: Iohexol
- Cohort 3: GFR: ≥ 30 and < 60 mL/min/1.73 m2 VFI dose: 47 mg/3 mL Number of doses: 1 Comparator: Iohexol 5 mL Comparator dose: 1
  Interventions: Device: VFI; Device: Iohexol
- Cohort 4: GFR: ≥ 15 and < 30 mL/min/1.73 m2 VFI dose: 47 mg/3 mL Number of doses: 1 Comparator: Iohexol 5 mL Comparator dose: 1
  Interventions: Device: VFI; Device: Iohexol

INTERVENTIONS:
Device: VFI — The IV administered visible fluorescent injectate (VFI)™ agent is comprised of a mixture of 2 different molecular weight carboxymethyl dextran molecules (5 kD and 150 kD) with different fluorescent dye molecules attached.
Device: Iohexol — Iohexol is a contrast enhancement agent which, following intravascular injection, is distributed in the extracellular fluid compartment and is excreted unchanged by glomerular filtration.
  Groups: Cohort 2; Cohort 3; Cohort 4

SUMMARY:
This is a Phase 2b, prospective, open-label study designed to evaluate the safety, tolerability, PK, and PD of FAST PV and mGFR Technology in healthy subjects and patients with varying degrees of renal impairment.

DETAILED DESCRIPTION:
For Cohorts 1 and 2, administration of the study drug will occur within 21 days of screening. Eligible subjects/patients will be admitted to the clinical research unit (CRU) on Day -1, at which time assessments will be performed, and results from both screening and Day -1 (inclusion/exclusion criteria, body weight, height [screening only], body mass index [BMI], medical and surgical history, physical examination, vital signs and pulse oximetry, 12 lead ECG, clinical laboratory tests, renal function assessment, follicle-stimulating hormone [FSH; screening only] and pregnancy test [females only], and urine drugs of abuse and alcohol screen) will be reviewed to confirm eligibility.

For Cohorts 3 and 4, administration of the study drug will occur within 21 days of screening. Eligible subjects/patients will be admitted to the CRU on Day 1, at which time assessments will be performed and results from both screening and predose administration testing (inclusion/exclusion criteria, body weight, height [screening only], BMI, medical and surgical history, physical examination, vital signs and pulse oximetry, 12 lead ECG, clinical laboratory tests, renal function assessment, FSH and pregnancy test [screening only], and urine drugs of abuse and alcohol screen) will be reviewed to confirm eligibility.

Cohort 1:

Eligible subjects will receive a single dose of VFI followed 130 minutes later by a 350 mL infusion of 5% albumin up to maximum volume of 7 mL/kg over 30 minutes on Day 1. Subjects will remain resident in the CRU for at least 24 hours after VFI administration for safety, PK, and PD assessments. Subjects will return to the CRU for an end-of-study (EOS) visit on Day 21 (± 1 day).

Cohort 2:

Eligible subjects will receive a dose of VFI followed 160 minutes later by a single dose of Iohexol on Day 1 and a second dose of VFI 24 hours following the initial dose of VFI. Subjects will remain resident in the CRU for at least 24 hours after the second VFI administration for safety, PK, and PD assessments. Subjects will return to the CRU for follow-up visits on Days 5 (± 1 day), 9 (± 1 day), and 16 (± 1 day) and an EOS visit on Day 22 (± 1 day).

Cohorts 3 and 4:

Eligible patients will receive a single dose of VFI followed 160 minutes later by a single dose of Iohexol on Day 1. Patients will remain in the CRU through the 12-hour sample collection after VFI administration for safety, PK, and PD assessments. . Patients will stay at a local hotel near the CRU and will return to the CRU on Day 2 for the 24-hour sample collection. Patients will return to the CRU for follow-up visits on Days 4 (± 1 day), 8 (± 1 day), and 15 (± 1 day) and an EOS visit on Day 21 (± 1 day).

ELIGIBILITY:
Inclusion Criteria:

All Subjects/Patients:

1. Males or females ≥ 18 and ≤ 75 years of age.
2. Females must be of non-childbearing potential (eg, postmenopausal [defined as cessation of regular menstrual periods for at least 1 year confirmed by follicle-stimulating hormone (FSH) test] or surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation [documentation required] or be using a medically acceptable form of birth control [eg, a barrier method, intrauterine device, or hormonal contraception]) from screening until 30 days after last dose.
3. Males who are sexually active and whose partners are females of childbearing potential must agree to practice abstinence or use condoms from screening through 90 days after administration of the last dose of study drug, and their partners must be willing to use a medically acceptable method of contraception (a barrier method, intrauterine device, or hormonal contraception) from screening through 90 days after administration of the last dose of study drug.
4. Males must agree to not donate sperm from screening through 90 days after administration of the last dose of study drug.
5. Subjects must be able to communicate effectively with the study personnel.
6. Subjects must be informed of the nature and risks of the study and give written informed consent prior to screening.
7. Body mass index ≥ 18.0 and ≤ 40.0 kg/m2, and body weight ≥ 40 kg at screening and CRU admission.

   BMI = weight (kg)/(height [m])2

   Subjects with Normal Renal Function (Cohorts 1 and 2):
8. Subjects must have an eGFR (calculated using the CKD-EPI Equation) ≥ 60 mL/min/1.73 m2 consistent with the National Kidney Foundation stages 1 and 2 of CKD.
9. Subjects must be otherwise healthy and without clinically significant abnormalities as assessed by review of medical and surgical history, physical examination, vital signs measurement, pulse oximetry, ECG, and clinical laboratory evaluations conducted at screening and CRU admission. A single repeat measurement/test may be performed, at the discretion of the physician, to confirm vital signs, pulse oximetry, ECG, and clinical laboratory tests abnormalities (ie, to confirm that a subject is eligible).

   Patients with Renal Impairment (Cohorts 3 and 4):
10. Patients in Cohort 3 must have an eGFR (calculated using the CKD-EPI Equation) ≥ 30 and < 60 mL/min/1.73 m2 consistent with the National Kidney Foundation stages 3a and 3b of CKD.
11. Patients in Cohort 4 must have an eGFR (calculated using the CKD-EPI Equation) ≥ 15 and < 30 mL/min/1.73 m2 consistent with the National Kidney Foundation stage 4 of CKD.
12. Patients may have clinical, ECG, and clinical laboratory findings consistent with their degree of renal dysfunction as assessed by review of medical and surgical history, physical examination, vital signs measurement, pulse oximetry, ECG, and clinical laboratory evaluations conducted at screening and CRU admission. A single repeat measurement/test may be performed, at the discretion of the physician, to confirm vital signs, pulse oximetry, ECG, and clinical laboratory tests abnormalities (ie, to confirm that a subject is eligible).

Exclusion Criteria:

All Subjects/Patients:

1. Female subject/patient is pregnant or breastfeeding.
2. History or presence of conditions which, in the judgment of the investigator, are known to interfere with the distribution, metabolism, or excretion of drugs.
3. History or presence of conditions that may place the subject at increased risk as determined by the investigator.
4. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
5. History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 6 months of screening.
6. Systolic blood pressure (BP) < 90 or > 160 mmHg or diastolic BP < 50 or > 100 mmHg measured after the subject has been resting quietly in a supine position or in the most recumbent position possible for at least 5 minutes at screening or CRU admission. A single repeat measurement may be performed to confirm vital signs abnormalities (ie, to confirm that a subject is eligible).
7. Heart rate (HR) < 40 or > 105 beats per minute (bpm) measured on ECG after the subject has been resting quietly in a supine position or in the most recumbent position possible for at least 5 minutes at screening or CRU admission. A single repeat measurement may be performed to confirm ECG abnormalities (ie, to confirm that a subject is eligible).
8. Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives of the investigational drug's PK, PD, or biological activity, whichever is longer, prior to first dose of study drug in this study.
9. Prior exposure to VFI or known allergy to dextrans.
10. History of any clinically significant allergic or negative reactions, side effects, or anaphylaxis to iodine, dyes, shellfish, isotopes, or dextran molecules.
11. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
12. Positive screen for human immunodeficiency virus (HIV)-1 or HIV-2 antibodies, hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
13. Diagnosis of acquired immune deficiency syndrome (AIDS).
14. History of nephrectomy or kidney transplant.
15. History of liver disease or screening liver function tests which exceed 2 × the upper limit of normal (ULN) or an albumin value of < 3 mg/dL.
16. International normalized ratio (INR) > 1.5 × ULN or a platelet count < 50,000.
17. Presence of significant hemodynamic instabilities.
18. Loss of Limb- as this alters the validity of eGFR and estimated PV equations.
19. Any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.
20. Involved in the planning or conduct of this study.
21. Inability to tolerate venipuncture or poor venous access.
22. Unwilling to abstain from alcohol from 24 hours prior to admission until discharge from the CRU.
23. Unwilling to abstain from strenuous activity (as assessed by the investigator) from 72 hours prior to admission until discharge from the CRU.
24. Unwilling or unlikely to comply with the requirements of the study.

    Subjects with Normal Renal Function (Cohorts 1 and 2):
25. Positive urine drugs of abuse or alcohol screen.
26. Use of prescription medications or any drugs that induce or inhibit study drug specific CYP(s) within 14 days or 5 half-lives, whichever is longer, of administration of the first dose of study drug.
27. Use of over the-counter (OTC) drugs (including herbal preparations) within 7 days or 5 half lives, whichever is longer, prior to administration of the first dose of study drug.

    Patients with Renal Impairment (Cohorts 3 and 4):
28. Clinically significant ongoing bleeding, changing hemoglobin, or experienced significant blood loss within 2 weeks prior to administration of the first dose of study drug.
29. Positive urine drugs of abuse (except for prescribed medications) or alcohol screen.
30. Use of anticoagulants and nonsteroidal anti-inflammatory drugs within 3 days prior to administration of the first dose of study drug.
31. Use of inotropes or vasopressors.
32. Any other condition or prior therapy that, in the investigator's opinion, is likely to deteriorate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) | 21 ± 1 days
  * Subjects will be monitored for AEs from administration of the first dose of study drug through the end of study visit
  * Abnormal clinical laboratory tests, physical examination findings, 12-lead electrocardiograms (ECGs), and vital signs including pulse oximetry that (1) are considered clinically significant initially and on confirmation, (2) require a subject to be discontinued from the study, (3) require a subject to receive treatment, or (4) require a change or discontinuation from the study drug (if applicable) will be recorded as AEs
Maximum observed plasma concentration (Cmax) | 21 ± 1 days
Time that Cmax was observed (tmax) | 21 ± 1 days
Area under the plasma concentration-time curve (AUC) from time 0 to 12 hours (AUC0 12: FD001 only) | 21 ± 1 days
AUC from time 0 to the time of the last quantifiable concentration (AUClast) | 21 ± 1 days
AUC from time 0 extrapolated to infinity (AUCinf) | 21 ± 1 days
Terminal elimination half-life (t½) | 21 ± 1 days
Terminal elimination rate constant (λz) | 21 ± 1 days
Total body clearance (CL) | 21 ± 1 days
Renal clearance (CLr; FD001 only) | 21 ± 1 days
Volume of distribution during the terminal phase (Vz) | 21 ± 1 days
Volume of distribution at steady state (Vss) | 21 ± 1 days
Fraction of dose excreted unchanged in the urine (Ae0-12) | 21 ± 1 days

SECONDARY OUTCOMES:
PV as assessed by FAST PV and mGFR Technology | 21 ± 1 days
PV as assessed by Nadler's formula | 21 ± 1 days
Changes in PV after fluid challenge | 21 ± 1 days
Repeatability of GFR measurements over 24 hours | 21 ± 1 days
mGFR as assessed by FAST VFI and Iohexol clearance methods | 21 ± 1 days
Estimated GFR (eGFR) (calculated by the Modification of Diet in Renal Disease [MDRD], Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] Creatinine and Cockcroft-Gault equations) | 21 ± 1 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DeNoia, MD, Principal Investigator — ICON Early Phase Services, LLC
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Division of Nephrology, Birmingham, Alabama
  - ICON Early Phase Services, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03095391/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03095391/SAP_001.pdf